CLINICAL TRIAL: NCT01625416
Title: Integrating Information Technology Advancements Into Early PTSD Interventions
Brief Title: Trauma Survivors Outcomes and Support Study IV
Acronym: TSOS IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001473; 1K24MH086814-01 (NIH); 1R01AA016102-01 (NIH)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Posttraumatic Stress Disorder; Depression; Suicide; Traumatic Brain Injury; Alcohol Use; Drug Use
Keywords: Posttraumatic Stress Disorder; Depression; Suicide; Traumatic Brain Injury; Alcohol Use; Drug Use; Information Technology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Suicide; Brain Injuries, Traumatic; Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped Care Management (Experimental): All patients randomized to receive the stepped care management procedures will meet with the trauma support specialist (TSS) prior to discharge from the hospital, who will provide coaching on use of mobile technology for mental health concerns. The TSS will complete follow-up correspondence across the 3-6 month time period to assess mental health functioning and use of information technology that addresses medical concerns. Patients who report barriers to mHealth technologies and request additional therapeutic services for mental health concerns assistance will receive evidence-based motivational interviewing and cognitive behavioral intervention procedures that can span up to 3-6 months.
  Interventions: Behavioral: Stepped Care Management
- Usual Care (No Intervention): Usual care control patients will be given a list of available community resources and encouraged to proceed using all resources available to them.

INTERVENTIONS:
Behavioral: Stepped Care Management — All patients randomized to receive the stepped care management procedures will meet with the trauma support specialist (TSS) prior to discharge from the hospital, who will provide coaching on use of mobile technology for mental health concerns. The TSS will complete follow-up correspondence across the 3-6 month time period to assess mental health functioning and use of information technology that addresses medical concerns. Patients who report barriers to mHealth technologies and request additional therapeutic services for mental health concerns assistance will receive evidence-based motivational interviewing and cognitive behavioral intervention procedures that can span up to 3-6 months.
  Arms: Stepped Care Management

SUMMARY:
After traumatic injuries some people have difficulty returning to the routine of their everyday activities and may experience physical and emotional pain. The purpose of this study is to identify new ways of providing support for physically injured trauma survivors. All study procedures are designed to work around patient needs and be as flexible as possible in order to best fit into patients' post-injury recovery.

Patients who are eligible for the study are randomly assigned to receive care as usual, or the "new method of treatment," with the study Trauma Support Specialist (TSS). This TSS will be in contact with the patient for the next three months; they may visit the patient at the hospital or at outpatient medical appointments. The TSS will also be available to talk with the patient over the telephone. Overall, the TSS will be working with the patient to help with difficulties returning to his or her routine and overcoming physical and emotional pain experienced after the injury. We believe that patients who receive the "new method of treatment," will be more able to return to daily routines and/or cope with the emotional stress that can occur after an injury. Intervention technology innovations including mHealth applications and web-based links will be included in the investigation.

DETAILED DESCRIPTION:
Clinical feasibility randomized clinical trial (RCT) pilot of integrating information technology advancements into Early PTSD Screening and Intervention. Design Overview: Between 30-200 injured trauma survivors who are initially admitted to either the Harborview inpatient wards or emergency department acute care settings will be enrolled in the study. If patients agree to participate, they will be engaged by a research assistant to complete a baseline assessment battery. Following the battery, all patients will be engaged in an initial technology readiness assessment to gauge comfort and skill using a variety of devices (e.g., smartphones, cellular phones, tablets, and laptop computers) that could potentially be utilized for delivery of interventions. Patients will then be randomized to either care as usual or to the stepped-care technology-based educational intervention. Patients randomized to the intervention condition will be met by a trauma support specialist. Intervention patients who endorse elevated substance use and/or mental health symptoms, including PTSD, depression, suicidal ideation, chronic pain, and postconcussive symptoms, will receive up to 3 months of motivational interviewing and/or cognitive behavioral therapy delivered by the trauma support specialist in person or over the telephone. The trauma support specialist may utilize mHealth technologies including websites and applications available on smartphones and tablet devices, as strategies to compliment CBT approaches that target specific areas of concern. However, the psychotherapeutic intervention embedded within the Stepped Care protocol is conceived of being fundamentally separate from the mHealth tools that may also be mentioned during discussions between the trauma support specialist and the patient. Inherent throughout the intervention is a focus on obtaining acceptability information from patients related to all aspects of the intervention and interpersonal experiences with the trauma support specialist, as well as any technology-based assessments and mHealth tools that may compliment the stepped care protocol. Patients will receive up to 3 consecutive months of trauma support specialist support post-injury. Follow-up assessments will occur at 1, 3, and 6 months following the baseline assessment, with additional acceptability assessments completed for specific aspects of the intervention listed above.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥3 on PTSD automated screening algorithm
* Score ≥35 on PTSD checklist (PCL-C)

Exclusion Criteria:

* Non-English speaking
* Under 14 years of age
* Patients in need of acute psychiatric intervention (e.g., suicide attempt, psychosis)
* Suffered head, spinal cord, or other sever injuries that prevent participation in the inpatient ward interview.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Zatzick, M.D., Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Zatzick D, O'Connor SS, Russo J, Wang J, Bush N, Love J, Peterson R, Ingraham L, Darnell D, Whiteside L, Van Eaton E. Technology-Enhanced Stepped Collaborative Care Targeting Posttraumatic Stress Disorder and Comorbidity After Injury: A Randomized Controlled Trial. J Trauma Stress. 2015 Oct;28(5):391-400. doi: 10.1002/jts.22041. PMID 26467327
- [Derived] Kelly CM, Van Eaton EG, Russo JE, Kelly VC, Jurkovich GJ, Darnell DA, Whiteside LK, Wang J, Parker LE, Payne TH, Mooney SD, Bush N, Zatzick DF. Technology Use, Preferences, and Capacity in Injured Patients at Risk for Posttraumatic Stress Disorder. Psychiatry. 2017 Fall;80(3):279-285. doi: 10.1080/00332747.2016.1271162. PMID 29087256

RESULTS

PARTICIPANT FLOW:
Groups:
- Stepped Care Management: Case management, information technology/mHealth innovations, psychotherapy, and psychopharmacology.: All patients randomized to receive the stepped care management procedures will meet with the trauma support specialist (TSS) prior to discharge from the hospital, who will provide coaching on use of mobile technology for mental health concerns. The TSS will complete follow-up correspondence across the three month time period to assess mental health functioning and use of information technology that addresses medical concerns. Patients who report barriers to mHealth technologies and request additional therapeutic services for mental health concerns assistance will receive evidence-based motivational interviewing and cognitive behavioral intervention procedures that can span up to 3-months.
Period: Overall Study
Arm/Group | Stepped Care Management | Usual Care
Started | 60 | 61
Completed | 51 | 54
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepped Care Management | Usual Care | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 57 | 112
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (14.7) | 43.5 (14.8) | 43.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 39 | 39 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 50 | 53 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 13 | 18
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 14 | 6 | 20
  White | 27 | 35 | 62
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Post Traumatic Stress Disorder (PTSD) Symptoms Over the Course of the Six Months After Injury
Description: The investigators used the PTSD Checklist - Civilian (PCL-C) as a continuous measure. The scoring of the scale ranges from a minimum of 17 to a maximum of 85, with higher scores indicating a worse outcome. No subscales were used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Management | Usual Care
Number analyzed (Participants) | 60 | 61
units on a scale
  Baseline | 47.0 (10.2) | 47.0 (10.9)
  1 month | 43.9 (16.1) | 43.6 (15.7)
  3 month | 41.4 (16.0) | 45.4 (16.0)
  6 month | 41.7 (16.2) | 47.1 (16.6)
Statistical Analysis 1: Comparison: Stepped Care Management vs Usual Care; Test type: Superiority; p = 0.05, Chi-squared; Chi square (2) =5.9, p=0.05; This chi-square analysis was derived from a mixed repeated measures model comparing intervention results with control results over 4 time points

2. Primary Outcome: Change in Depression Symptoms Over the Course of the Six Months After Injury
Description: The investigators used the Patient Health Questionnaire (PHQ-9) as a continuous measure, with scores ranging from 1 to 27. Higher scores represent a worse outcome. No subscales were used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Management | Usual Care
Number analyzed (Participants) | 60 | 61
units on a scale
  Baseline | 14.3 (5.7) | 15.0 (5.0)
  1 month | 13.2 (6.3) | 13.8 (6.1)
  3 month | 12.5 (6.4) | 14.1 (7.4)
  6 month | 12.5 (7.2) | 14.4 (7.2)
Statistical Analysis 1: Comparison: Stepped Care Management vs Usual Care; Test type: Superiority; p = 0.69, Chi-squared; Chi square(2) = 0.74, p = 0.69; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Technology Use
Description: The investigators used laptop tracking software to determine technology usage.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Stepped Care Management | Usual Care
Number analyzed (Participants) | 60 | 61
minutes | 24.76 (42.51) | 16.05 (26.82)

4. Primary Outcome: Feasibility/Acceptability of Intervention
Description: The investigators used laptop tracking software to assess number of patients using laptops.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Care Management | Usual Care
Number analyzed (Participants) | 60 | 61
Participants | 37 | 33

5. Secondary Outcome: Alcohol Use Problems
Description: The investigators used the Alcohol Use Disorders Identification Test (AUDIT) as a continuous measure. The 10-item scale score ranges from 0-40, with higher values indicating a worse outcome. No sub scales were used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Management | Usual Care
Number analyzed (Participants) | 60 | 61
units on a scale
  Baseline | 4.5 (3.4) | 4.2 (3.9)
  1 month | 1.5 (2.7) | 1.0 (2.3)
  3 month | 2.4 (3.1) | 1.9 (3.1)
  6 month | 2.7 (3.0) | 2.1 (2.8)
Statistical Analysis 1: Comparison: Stepped Care Management vs Usual Care; Test type: Superiority; p = 0.97, Chi-squared — Chi square (2) = 0.06, p = 0.97; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Physical Functioning
Description: The investigators used the Medical Outcomes Study Short Form healthy survey (MOS SF-12/36) physical components summary to assess physical function. The minimum and maximum scores are 0-100 with higher scores representing a better outcome. No other subscales will be used.
Time Frame: The investigators assessed at baseline, 1-, 3-, and 6-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Care Management | Usual Care
Number analyzed (Participants) | 60 | 61
units on a scale
  Baseline | 47.3 (13.0) | 42.8 (14.0)
  1 month | 27.9 (11.8) | 27.4 (11.6)
  3 month | 35.2 (13.1) | 33.6 (13.4)
  6 month | 36.9 (11.5) | 34.6 (12.3)
Statistical Analysis 1: Comparison: Stepped Care Management vs Usual Care; Test type: Superiority; p = 0.71, Chi-squared; Chi-Square (2) =0.68, p=0.71; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Stepped Care Management | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 31/60 | 36/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stepped Care Management (N=60) | Usual Care (N=61)
Suicide ideation (Psychiatric disorders) | 31 | 36 — PHQ-9 Score of >0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No